CLINICAL TRIAL: NCT00591799
Title: Clinical Protocol for Evaluation of the Jarvik 2000 Heart Assist System
Brief Title: Jarvik 2000 Heart as a Bridge to Cardiac Transplantation - Pivotal Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jarvik Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G000058
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Jarvik 2000 Ventricular Assist System (Experimental): Jarvik 2000 Ventricular Assist System
  Interventions: Device: The Jarvik 2000 Ventricular Assist System

INTERVENTIONS:
Device: The Jarvik 2000 Ventricular Assist System — Jarvik 2000 Heart implantation is intended for patient's with end-stage heart failure who are approved heart transplant candidates - who meet all of the study's inclusion criteria and none of its exclusion criteria.
  Other Names: Jarvik 2000

SUMMARY:
The purpose of the study is to determine the safety and effectiveness of the Jarvik 2000 Heart as a bridge to heart transplantation in end-stage heart failure patients who are approved heart transplant candidates.

DETAILED DESCRIPTION:
The Jarvik 2000 Heart is a silent compact axial flow impeller pump of 1 inch diameter, weighing 90g with a displacement volume of 25ml. The pump is implanted into the apex of the left ventricle by left thoracotomy, or by mid-sternotomy, or by the subcostal approach. A vascular graft offloads to either the descending thoracic aorta, the ascending thoracic aorta, or the abdominal aorta. The impeller rotates at speeds of 8,000 to 12,000 rpm providing blood flow of up to seven L/minute. At higher speeds the pump can produce 10 L/minute. Power is provided through an abdominal drive line.

ELIGIBILITY:
Inclusion Criteria: (The following are general inclusion criteria; more specific criteria are outlined in the study protocol).

* Transplant listed UNOS status IA or IB patients.
* BSA >1.5 m2 and <2.3 m2.
* Dependent on one or more intravenous inotropic agents or an intraaortic balloon pump (IABP).

Exclusion Criteria:(The following are general exclusion criteria; more specific criteria are outlined in the study protocol).

* Known risk factors or conditions that would contraindicate LVAD implantation or adversely affect patient survival.
* Evidence of end organ dysfunction.
* Known coagulopathy or contraindication of anticoagulation or antiplatelet agents.
* Systemic infection.
* Malignancies not in remission.
* Current participation in investigational trials with other devices, drugs, or biologic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Survival to cardiac transplantation or survival and transplant listed at 180 days following implant of the Jarvik 2000 Heart. | 180 days

SECONDARY OUTCOMES:
Incidence of serious adverse events as events per patient month including infection, stroke, VAD failure, and all serious adverse events. Quality of Life measures - MLHFQ, NYHA class, Neurocognitive assessments. | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jarvik, MD, Study Chair — Jarvik Heart, Inc. SPONSOR
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Selzman CH, Feller ED, Walker JC, Sheridan BC, Silvestry SC, Daly RC, Anyanwu AC, Madigan D, Liu PY, Frazier OH, Jorde UP, Griffith BP. The Jarvik 2000 Left Ventricular Assist Device: Results of the United States Bridge to Transplant Trial. ASAIO J. 2023 Feb 1;69(2):174-182. doi: 10.1097/MAT.0000000000001750. Epub 2022 Apr 13. PMID 35421002